CLINICAL TRIAL: NCT06498635
Title: Randomized Phase III Trial INcorporating Pathologic Complete ReSponse in Participants With Early StaGe Non Small Cell Lung Cancer to Optimize ImmunotHerapy in The AdjuvanT Setting (INSIGHT)
Brief Title: Immunotherapy After Surgery for People Who Have No Remaining Cancer Cells After Standard Treatment for Early-Stage Non-Small Cell Lung Cancer, INSIGHT Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-05588; NCI-2024-05588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2414 (Other: SWOG); S2414 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2024-07-10; First posted 2024-07-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; durvalumab; Immunoglobulin G; Disulfides; Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (durvalumab) (Experimental): Patients receive durvalumab IV over 60 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT and blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Other: Questionnaire Administration
- Arm II (active surveillance) (Active Comparator): Patients undergo active surveillance for 12 months on study. Patients undergo CT and blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Patient Observation; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
  Arms: Arm I (durvalumab)
Other: Patient Observation — Undergo active surveillance
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Arm II (active surveillance)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares durvalumab to the usual approach (patient observation) after surgery for the treatment of patients with early-stage non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The usual approach for patients who are not in a study is to closely watch a patient's condition after surgery and to have regular visits with their doctor to watch for signs of the cancer coming back. Usually, patients do not receive further treatment unless the cancer returns. This study will help determine whether this different approach with durvalumab is better, the same, or worse than the usual approach of observation. Giving durvalumab may help patients live longer and prevent early-stage non-small cell lung cancer from coming back as compared to the usual approach.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare disease free survival (DFS) in stage II-IIIB non-small cell lung cancer participants who achieved a pathologic complete response (pCR) following standard of care neoadjuvant chemo-immunotherapy and are randomized to adjuvant durvalumab (MEDI4736) versus surveillance.

SECONDARY OBJECTIVES:

I. To compare the overall survival (OS) between the arms. II. To evaluate the frequency and severity of toxicities of adjuvant durvalumab (MEDI4736).

III. To compare the event free survival (EFS) between the arms.

TRANSLATIONAL MEDICINE OBJECTIVE:

I. To bank specimens and images for additional future translational medicine studies.

QUALITY OF LIFE (QOL) PRIMARY OBJECTIVE:

I. To compare patient-reported quality of life (QOL) status between treatment arms at 6 months from randomization using the Functional Assessment of Cancer Therapy-Lung (FACT-L) Trial Outcome Index (TOI).

QOL SECONDARY OBJECTIVES:

I. To compare patient-reported QOL between treatment arms at 24 weeks (6 months) from randomization using the Functional Assessment of Cancer Therapy-Biologic Response Modifier (FACT-BRM) physical and mental subscale scores.

II. To compare longitudinal changes in global health status between treatment arms from randomization to 48 week (12 months) using the FACT-L TOI.

PATIENT REPORTED OUTCOMES-COMMON TERMINOLOGY CRITERIA FOR ADVERSE EVENTS (PRO-CTCAE) OBJECTIVE:

I. To compare participant-reported symptoms using selected PRO-CTCAE items between treatment arms such as rash, itching, skin dryness, numbness, and tingling.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive durvalumab intravenously (IV) over 60 minutes on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) and blood sample collection throughout the trial.

ARM II: Patients undergo active surveillance for 12 months on study. Patients undergo CT and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up annually until 10 years from randomization.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytological confirmed diagnosis of clinical stage II-IIIB (excluding clinical N3 disease) non-small cell lung cancer (NSCLC)
* Participants must have had a complete (R0) resection of NSCLC (with appropriate lymph node sampling as defined by the National Comprehensive Cancer Network [NCCN] guidelines) within 84 days (12 weeks) prior to randomization. Acceptable types of surgical resection are: lobectomy, sleeve resection, bi-lobectomy, or pneumonectomy. Wedge resection is not allowed.

  * Note the NCCN guidelines: N1 and N2 node resection and mapping is a routine component of lung cancer resections. It is recommended at a minimum one N1 and three N2 stations is sampled or complete lymph node dissection. Formal ipsilateral mediastinal lymph node dissection is indicated for participants undergoing resection for N2 disease
* Participants must have a pathologic complete response (pCR) (no viable tumor in the resected specimen or lymph nodes), as determined by local pathology review
* Participants must have a PD-L1 status result (e.g. [< 1% versus >= 1% or unknown])
* Participants must not have known EGFR mutations, or ALK gene fusion
* Participants must have received at least two cycles of neoadjuvant platinum-based chemotherapy and anti-PD-1 or anti-PD-L1 therapy. The neoadjuvant treatment must be Food and Drug Administration (FDA) approved and standard of care as listed in NCCN guidelines
* Participants must not be planning to receive any concurrent non-protocol directed chemotherapy, immunotherapy, biologic or hormonal therapy for NSCLC treatment while receiving treatment on this study
* Participants must not have received any prior systemic therapy (systemic chemotherapy, immunotherapy or investigational drug) within 28 days prior to randomization
* Participants must not have medical contraindications or severe adverse events to receiving anti-PD-1 or anti-PD-L1 therapy
* Participants must not have received post-operative radiation therapy (PORT) for NSCLC
* Participants must not have any unresolved toxicity National Cancer Institute (NCI) CTCAE grade ≥ 2 from previous anticancer therapy with the exception of alopecia, and vitiligo. Note, participants with grade ≥2 neuropathy may be included at the discretion of the treating investigator. Note, participants with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included at the discretion of the treating investigator
* Participant must be ≥ 18 years old at time of study entry
* Participants must have body weight > 30 kg
* Participant must have Zubrod performance status of 0-2
* Participant must have a complete medical history and physical exam within 28 days prior to randomization
* Hemoglobin > 9.0 g/dL (within 28 days prior to randomization)
* Absolute neutrophil count ≥ 1.5 x 10^3/uL (within 28 days prior to randomization)
* Platelets ≥ 100 x 10^3/uL (within 28 days prior to randomization)
* Total bilirubin ≤ 1 x institutional upper limit of normal (ULN) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin ≤ 5 x institutional ULN (within 28 days prior to randomization)
* Aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 3 × institutional ULN (within 28 days prior to randomization)
* Participants must have a calculated creatinine clearance ≥ 40 mL/min using the following Cockcroft-Gault formula. This specimen must have been drawn and processed within 28 days prior to randomization. For creatinine clearance formula see the tools on the Clinical Research Associate (CRA) Workbench https://txwb.crab.org/TXWB/Tools.aspx
* Participants must have fully recovered from the effects of prior surgery in the opinion of the treating investigator
* Participants with a known history of human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at registration and have undetectable viral load test on the most recent test results obtained within 6 months prior to randomization
* Participants with a known history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load while on suppressive therapy on the most recent test results obtained within 6 months prior to randomization, if indicated
* Participants with a known history of hepatitis C virus (HCV) infection must have been treated and cured. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 6 months prior to randomization, if indicated
* Participants must not have had an organ transplant
* Participants must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participant must not have medical contraindications to receiving immunotherapy, including history of non-infectious pneumonitis that required steroids or active autoimmune disease that has required systemic treatment with disease modifying agents, corticosteroids or immunosuppressive drugs in the past two years. Replacement therapy (e.g. thyroxine for pre-existing hypothyroidism, insulin for type I diabetes mellitus, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Intra-articular steroid injections are allowed
* Participants must not be pregnant or nursing (nursing includes breast milk fed to an infant by any means, including from the breast, milk expressed by hand, or pumped). Individuals who are of reproductive potential must have agreed to use an effective contraceptive method during protocol therapy and for 6 months following completion of protocol therapy with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen. Participants should not breastfeed during protocol therapy and for 6 months following completion of protocol therapy
* Participants must not have received a live or live attenuated vaccine within 28 days prior randomization. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever rabies, Bacillus Calmette-Guerin (BCG) and typhoid vaccine. Seasonal influenza vaccines and coronavirus disease 19 (COVID-19) vaccines are allowed, however, intranasal influenza vaccines (e.g. Flu-Mist) are live attenuated, and are not allowed
* Participants must be offered the opportunity to participate in specimen banking
* Participants who can complete FACT-L, FACT-BRM, and PRO-CTCAE questionnaires forms in English, or Spanish must agree to participate in the patient-reported outcome study
* NOTE: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines
* For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2039-07-15 (Estimated); Study Completion 2039-07-15 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | From date of randomization to the earliest event defined as date of first documentation of recurrence, any new lung cancer (even in the contralateral lung), or death due to any cause, assessed up to 10 years
  Will be assessed using a 1-sided 5% level log-rank test accounting for interim testing, stratified on the randomization stratification factors.

SECONDARY OUTCOMES:
Event-free survival (EFS) | From date of randomization to date of first occurrence of EFS event, assessed up to 10 years
  EFS events are defined as: Discontinuation of durvalumab (MEDI4736) due to toxicity, either immune or non-immune related, any new lung cancer (even in the contralateral lung), the use of glucocorticoids for > 14 days for the treatment of toxicity secondary to durvalumab (MEDI4736), hospitalization due to toxicity from durvalumab (MEDI4736), disease recurrence, or death due to any cause. Will be estimated using the method of Kaplan-Meier. 95% confidence for the medians will be constructed using the method of Brookmeyer-Crowley. Hazard ratios (HRs) and corresponding 90% confidence intervals (CI) will be estimated using a Cox proportional hazards model with treatment arm as a single covariate. EFS will be compared between treatment arms using log-rank test, stratified on the randomization stratification factors.
Overall survival (OS) | From date of randomization to date of death due to any cause, assessed up to 10 years
  Will be estimated using the method of Kaplan-Meier. 95% confidence for the medians will be constructed using the method of Brookmeyer-Crowley. HRs and corresponding 90% CI will be estimated using a Cox proportional hazards model with treatment arm as a single covariate. OS will be compared between treatment arms using log-rank test, stratified on the randomization stratification factors.
Incidence of adverse events | Up to 10 years
  Will be evaluated using the Common Terminology Criteria for Adverse Events version 5 items. Binary proportions and associated confidence intervals will be calculated.

OTHER OUTCOMES:
Patient reported outcomes | Up to 10 years
  Will be assessed by Patient Reported Outcomes - Common Terminology Criteria for Adverse Events (PRO-CTCAE) instrument(s). For each of the PRO-CTCAE adverse events examined, the scores for each attribute (frequency, severity and/or interference) will be presented descriptively using summary statistics at each assessment time. Additionally, the worst severity and/or interference over the entire course will be summarized.
Estimates of the primary outcome treatment effect | Up to 10 years
  The hazard ratio of DFS and the corresponding 95% CIs will be estimated for subgroups defined by sex, race and ethnicity, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy P Cetnar, Principal Investigator — SWOG Cancer Research Network
Locations (209):
- United States (209):
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Hartford HealthCare - Avon, Avon, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Hartford HealthCare - Manchester, Manchester, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Northwestern Medicine Huntley Hospital, Huntley, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - UPMC Western Maryland, Cumberland, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Duke Cancer Center Cary, Cary, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Hood River Memorial Hospital, Hood River, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm